CLINICAL TRIAL: NCT05634460
Title: Comparison of 5% Potassium Hydroxide With 10% Potassium Hydroxide Solution in Treatment of Molluscum Contagiosum
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Combined Military Hospital Abbottabad (Other)
Responsible Party: Principal Investigator, Huma Farid, Dr. Huma Farid, Combined Military Hospital Abbottabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMHAtd-ETH-04-Derm-22
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Molluscum Contagiosum
Keywords: potassium hydroxide 5% and 10% lotion
MeSH Terms: conditions — Molluscum Contagiosum | interventions — potassium hydroxide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): patients in group A treated with 5% potassium hydroxide on every lesion once daily via cotton-tipped applicator for at least two weeks or till inflammatory manifestations
  Interventions: Drug: potassium hydroxide
- group B (Active Comparator): patients in group B treated with10% potassium hydroxide on every lesion once daily via cotton-tipped applicator for at least two weeks or till inflammatory manifestations
  Interventions: Drug: potassium hydroxide

INTERVENTIONS:
Drug: potassium hydroxide — Potassium hydroxide (KOH) is a topical treatment for Molluscum contagiosum. Dermatologists routinely use potassium hydroxide (KOH) in varying concentrations to identify fungal elements. Because it is a strong alkali with keratolytic characteristics, variable concentrations given for management of MC.

SUMMARY:
Molluscum is a virus-related skin infestation which is commonly seen among children. Molluscipox virus, the largest human virus, causes it. MC typically manifests as a single or multiple dome-shaped, shiny, pearly white papules with a central dimple. In immunocompetent individuals, spontaneous resolution usually occurs within 18 months; however, the lesion may persist for several years. Asymptomatic lesions are common. It is also linked to a high risk of transmission and an increasing prevalence in global populations1-2.

Patients may receive therapy for social and cosmetic reasons, and also to avoid spreading disease to others. Numerous modalities are currently available, including Potassium hydroxide, curettage, cryotherapy, disinfected needle pricking, photodynamic therapy, laser, salicylic acid, glycolic acid etc3-4.

Potassium hydroxide (KOH) is a topical treatment for Molluscum contagiosum. Dermatologists routinely use potassium hydroxide (KOH) in varying concentrations to identify fungal elements. Because it is a strong alkali with keratolytic characteristics, variable concentrations given for management of MC. Because it is inexpensive and widely accessible, it has the potential to be a useful method for treating for MC in resource-constrained countries5-6.

The purpose of this study is to examine two varied concentrations of Potassium hydroxide (5%-KOH vs 10%-KOH) among MC patients in order to determine the most effective KOH concentration to manage Molluscum Contagiosum among children.

ELIGIBILITY:
Inclusion Criteria <100 lesions no therapy within the earlier one month

Exclusion Criteria:

known hypersensitivity and immunodeficiency

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
. Efficacy was classified as follows: • complete remission (≥ 90% clearance of lesions) • partial remission (60-90% clearance of lesions) • insignificant improvement (<60% clearance of lesions) | 06 months

CONTACTS AND LOCATIONS:
Overall Officials: Bushra Muzaffar, FCPS, Principal Investigator — Combined Military Hospital Abbottabad
Locations (1):
- CMH, Abbottabad, KPK, Pakistan